CLINICAL TRIAL: NCT06695507
Title: Upfront Ruxolitinib Treatment for Chronic Graft-vs-host Disease in Children and Young Adults: A Corticosteroid-sparing Pilot Study
Brief Title: Upfront Ruxolitinib for Chronic Graft-vs-host Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0529
Record Dates: First submitted 2024-11-16; First posted 2024-11-19 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib Treatment (Experimental)
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Participants will receive ruxolitinib for 6 months.

SUMMARY:
While hematopoietic stem cell transplant (HSCT) is an effective therapy, graft versus host disease (GVHD) is the most significant complication after HSCT. Corticosteroids (or steroids) have been the mainstay of treatment for chronic GVHD for many decades now. Increasingly, newer immunosuppressive and immunomodulating agents are being studied in adults and children affected by cGVHD. Ruxolitinib is one of these promising newer agents, which has been shown to be effective in the treatment of cGVHD in both children and adults. Currently, ruxolitinib is generally added to a patient's treatment regimen after (or with) a course of high dose steroids.

The purpose of this study is to examine the effectiveness of upfront single agent ruxolitinib for cGVHD.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed moderate to severe chronic graft versus host disease (as defined by NIH cGVHD consensus criteria), requiring systemic treatment
* Patient aged ≥12 year-old and ≤30 year-old
* Patient able to take oral or enteral medication
* No active, clinically significant uncontrolled infections
* ALT ≤ 5x upper limit of normal (ULN) and total bilirubin ≤ 5xULN (unless presumed liver GVHD)
* Platelet ≥ 20k and ANC ≥ 500. The use of transfusions or growth factors is permitted to maintain counts at these thresholds
* No prior systemic treatment for chronic GVHD. Patients previously treated for acute GVHD are eligible, including those who received ruxolitinib for treatment of their aGVHD
* Patients must be on ≤ physiologic dosing (i.e. hydrocortisone 8-12mg/m2/day) at enrollment
* Patients with prior acute GVHD on < 1 mg/kg steroids with new onset moderate-severe chronic GVHD may be considered for enrollment if they can taper steroids to reach physiological hydrocortisone in 1 month. If unable to do so these patients will come off study and be replaced

Exclusion Criteria:

* Mild cGVHD (as defined by NIH cGVHD consensus criteria11), that does not require systemic therapy
* Acute or late acute GVHD without any evidence of chronic GVHD features
* Patients who have received corticosteroids for ≥ 24 hours at 1 mg/kg/day of methylprednisolone or prednisone with the intent to treat cGVHD at time of enrollment
* Corticosteroid dosing above physiologic dose hydrocortisone (i.e. > 8-12mg/m2/day) at time of enrollment
* Clinical evidence suggesting active malignancy (including PTLD and primary/secondary malignancy)
* Clinical evidence of clinically significant active infection
* Ongoing cytopenias which cannot be supported with routine supportive care (keeping hemoglobin over 7 g/dL and platelets >20,000 and absolute neutrophil count over 500/uL)
* Active lower gastrointestinal bleeding
* Thrombosis within 6 months (including myocardial infarction, stroke, deep venous thrombosis, pulmonary embolism). IV infiltration will not be included as an example of thrombosis
* Pregnant or lactating females; patients of childbearing age who are not able to comply with contraceptive recommendations
* Other condition that PI feels would preclude the patient from complying with study activities
* ESRD [CLcr < 15 mL/min] not on dialysis
* Overlap syndrome

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Khandelwal, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States